CLINICAL TRIAL: NCT06661369
Title: Comparative Effects of Individual and Grouped Sensory Perceptual Motor Training on Gross Motor Skills and Quality of Life in Children With Autism Spectrum Disorder
Brief Title: Study Comparing the Effects of SPM Techniques, Individually vs. Grouped in Children With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/Sara Sattar
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; sensory perceptual motor training; Test of Movement Battery for children,; DSM-5
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial in which non probability convenient sampling will be used. Two groups of 4-12 age will be formed in which participants will be randomly divided. Group A: individually SPM training will be given, Group B: Grouped SPM training given
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual ASD Children (Experimental): Activities were applied individually for the IND group. Individual training was applied according to the treatment protocol, activities done by step by step from simple to complex. Each activities for individuals training will be applied for 2 hours, three sessions per week, for ten successive months
  Interventions: Other: Sensory Perceptual Motor Training on Individual
- Group of ASD Children (Experimental): Activities were applied in group . Group training was applied according to the treatment protocol, activities done by step by step from simple to complex. each activities for group training will be applied for 2 hours, three sessions per week, for ten successive months
  Interventions: Other: Sensory Perceptual Motor Training on Group

INTERVENTIONS:
Other: Sensory Perceptual Motor Training on Group — 1. Sensory Input
     * Wheelbarrow walks, swimming, and drying off.
  2. Proprioceptive
     * Climbing, pushing, pulling, and carrying heavy objects.
  3. Vestibular
     * Swinging, trampolining, and playground games.
  4. Tactile
     * Stereognosis training, textured paths, and messy play (mud, sand).
  5. Motor Planning
     * Statue spinning, crawling through/under objects, and quick movements.
  6. Balance and Posture
     * Various balance positions (e.g., hands and knees).
  7. Ocular Control
     * Catching and tossing balls.
  8. Bilateral Coordination
     * Activities using both sides of the body (e.g., stick ball).
  9. Visual-Spatial
     * Walking, stair climbing, and puzzles.
  10. Fine Motor Skills
      * Puzzles, bead stringing, and drawing.
  11. Gross Motor
      * Standing, walking, running, and throwing games.
  Arms: Group of ASD Children
Other: Sensory Perceptual Motor Training on Individual — 1. Sensory Input
     * Wheelbarrow walks, swimming, and drying off.
  2. Proprioceptive
     * Climbing, pushing, pulling, and carrying heavy objects.
  3. Vestibular
     * Swinging, trampolining, and playground games.
  4. Tactile
     * Stereognosis training, textured paths, and messy play (mud, sand).
  5. Motor Planning
     * Statue spinning, crawling through/under objects, and quick movements.
  6. Balance and Posture
     * Various balance positions (e.g., hands and knees).
  7. Ocular Control
     * Catching and tossing balls.
  8. Bilateral Coordination
     * Activities using both sides of the body (e.g., stick ball).
  9. Visual-Spatial
     * Walking, stair climbing, and puzzles.
  10. Fine Motor Skills
      * Puzzles, bead stringing, and drawing.
  11. Gross Motor
      * Standing, walking, running, and throwing games.
  Arms: Individual ASD Children

SUMMARY:
Autism is the most prevalent disorder as it affects attention, awareness, cognitive development, social development, and emotional aspects too. It is one of the comprehensive developmental disorders in the early stage, which is characterized by weak social learning and communication, limited activities, interests, learning, insufficient imaginative and stereotypical thinking or non-functional thinking of movements and verbalities. A lack of sensory perception leads to a leading autistic child's sensitivity to sensory stimuli or weak sensitivity and the child is not aware of the surrounding environment.

DETAILED DESCRIPTION:
The current study will be randomized control trial; data will be collected from Lahore Garrison Institute of Special Education. This study will be conducted with 32 participants equally divided into two groups. Inclusion criteria will be Children who diagnosed with Autism Spectrum Disorder (mild & moderate) according to Diagnostic and Statistical Manual of Mental Disorders, (DSM-5), Have an IQ 70 according to Stanford-Binet Intelligence Scales and be able to understand and follow instructions, Children whose age between 4 to 12 and All participants had to be able to sit and walk without support according to GMFCS. Exclusion criteria for the study include Children who will associate with attention deficit hyperactivity disorder signs, Upper limb musculoskeletal injuries, Visual or auditory impairments, Children who had received sensory integration therapy for > 3 months within the past 6 months and Children with speech delay, hearing impairment, or intellectual disability. SPM training will be given each child individually in the first group. In the second group techniques will be apply in a group therapy. The SPM training programme will apply for 10 months. Outcomes, including the Test of Movement Battery for Children, Quality of life scale will be use. Data analysis will be performed using SPSS version 23.00

ELIGIBILITY:
Inclusion Criteria:

* Children who diagnosed with Autism Spectrum Disorder (mild & moderate) according to Diagnostic and Statistical Manual of Mental Disorders, (DSM-5)
* Have an IQ 70 according to Stanford-Binet Intelligence Scales
* Children whose age between 4 to 12
* All participants had to be able to sit and walk without support

Exclusion Criteria:

* Children who will associate with attention deficit hyperactivity disorder signs
* Upper limb musculoskeletal injuries
* Visual or auditory impairments
* Children who had received sensory integration therapy for > 3 months within the past 6 months
* Children with speech delay, hearing impairment, or intellectual disability

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
THE DEVELOPMENTAL COORDINATION The Developmental Coordination Disorder Questionnaire | 10-15 minutes
  The Developmental Coordination Disorder Questionnaire (DCDQ) is a parent-report screening tool for identifying motor coordination difficulties in children aged 5 to 15 years, 11 months. It includes 15 items across three domains: Control During Movement, Fine Motor/Handwriting, and General Coordination, rated on a 5-point Likert scale. Scores below age-specific cutoffs suggest potential Developmental Coordination Disorder (DCD). It is reliable, quick (10-15 min), but not diagnostic, requiring further evaluation.

SECONDARY OUTCOMES:
Short Sensory Profile | 2-5 hours
  The Short Sensory Profile (SSP) is a caregiver-completed questionnaire used to assess sensory processing difficulties in children aged 3-14 years. It includes 38 items across seven domains (e.g., tactile sensitivity, auditory filtering), rated on a 5-point scale. Scores help identify sensory modulation issues affecting daily activities. The SSP is quick, reliable, and widely used, but it is a screening tool, not a diagnostic instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Sattar, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No